CLINICAL TRIAL: NCT03134430
Title: Effects of Regional Nerve Block on Cancer Recurrence
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Luo Foquan (Other)
Responsible Party: Sponsor-Investigator, Luo Foquan, Professor, The First Affiliated Hospital of Nanchang University
Organization: The First Affiliated Hospital of Nanchang University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LFoquan
Record Dates: First submitted 2017-03-20; First posted 2017-05-01 (Actual); Last update posted 2018-05-25 (Actual); Status verified 2018-05

CONDITIONS: Cancer Patient
Keywords: Regional nerve block; cancer recurrence
MeSH Terms: interventions — Saline Solution

STUDY DESIGN:
Intervention Model Description: the patients in treatment group will received reginoal nerve block with 0.35% Ropivacane and 0.5% lidocaine in normal saline under ultrasound guide, while those in control group received equal volume of normal saline.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Normal saline (Placebo Comparator): equal volume of normal saline as treatment group
  Interventions: Other: Normal saline
- peripheral Nerve block (Active Comparator): 0.35% ropivacaine and 0.5% lidocaine in normal saline
  Interventions: Other: peripheral Nerve block

INTERVENTIONS:
Other: Normal saline — Injection of Normal saline around peripheral nerve
  Arms: Normal saline
Other: peripheral Nerve block — Injection of local anesthetics around peripheral nerve
  Arms: peripheral Nerve block

SUMMARY:
It has been reported local anesthetics could inhibit tumor cell proliferation, metastasis and invasion ability，but it is still lack of clinical evidence. Our study aims to explore the effects of regional nerve block on cancer recurrence and the mechanism.

DETAILED DESCRIPTION:
1. To study the effects of TAP block under ultrasound guide on the recurrence of gastric carcinoma, colon cancer, rectal carcinoma and liver cancer and the underlying mechanisms.
2. To clarify the effects of Lateral thoracic nerve block under ultrasound guide on the recurrence of lung cancer and the underlying mechanisms.

ELIGIBILITY:
Inclusion Criteria:

* Patients with primary cancer undergoing elective surgery under general anesthesia

Exclusion Criteria:

* Disagree to participate，drop out,lose track, infectious abdominal wall，abnormal puncture point，coagulation dysfunction，allergy of local anesthetic ，immune disease,cancer metastasis,mental disease, acute and chronic infectious disease or other severe disease.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2017-07-10 (Actual); Primary Completion 2018-03-25 (Actual); Study Completion 2023-05-01 (Estimated)

PRIMARY OUTCOMES:
the effect of nerve block on the cancer recurrence rate and survival rate postoperation | up to 5 years after surgery
  to trace cancer recurrence after tumor resection with CT scaning and tumor biological maker test for 5 years

SECONDARY OUTCOMES:
dosage of intraoperative anesthetic | intraoperative period
  Record the propofol and remifentanil during the operation
the effect of nerve block on the percentage and classification of immunocyte and content of cytokines | at 0h, 24h, 48h after nerve block
  percentage and classification of immunocyte will be detected by Use flow cytometry, and cytokines will be detected by ELISA
VAS after operation | at 24h, 48h after nerve block
  Assess the visual analogue scale 24，48h after nerve block
activity after operation | up to 2 weeks
  Observe recovery time of gastrointestinal function and off-bed activity after nerve block
Hospital stay | up to 4 weeks after surgery
  Observe length of hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Foquan Luo, professor, Study Chair — The First Affiliated Hospital of Nanchang University
Locations (1):
- The first affiliated hospital of nanchang university, Nanchang, Jiangxi, China